CLINICAL TRIAL: NCT05472675
Title: Local Sensory Nerve Block in the Treatment of Vestibular Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Head of Department of Otolaryngology, Pamukkale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2022-07-14; First posted 2022-07-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Vestibular Migraine
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- local anesthetic and botulinum toxin group (Experimental): patients who have vestibular migraine and who accepted for study gruoup as local anesthetic and botulinum toxin group
  Interventions: Procedure: Botulinum toxin and bupivacain

INTERVENTIONS:
Procedure: Botulinum toxin and bupivacain — Botulinum toxin A AND bupivacain( local anesthetic)

SUMMARY:
There is no standard approach to the treatment of vestibular migraine. Agents used in the treatment of migraine are frequently used. In treating migraine, local anesthetic agents, nerve-blocking methods, and botulinum toxin local injection is commonly applied, and successful results are obtained. Adapting the nerve-blocking method used in the treatment of migraine to the treatment of vestibular migraine is the purpose of the study.

DETAILED DESCRIPTION:
Patients between 18-75 diagnosed with/without aura or chronic migraine according to IHCD-3 diagnostic criteria and who describe dizziness during or between attacks will be evaluated in the ENT clinic.

Patients included in the study will be recorded as definite vestibular migraine or probable vestibular migraine according to criteria defined in the BARANY community and IHCD-3. Differential diagnosis of vertigo will be made with pure tone audiometry, Caloric test, VHIT, Videonystagmography, and cVEMP. MIDAS (migraine disability scale), DHI (dizziness handicap inventory), VSS (vertigo symptom scale), DASÖ-21 anxiety test, and Allodynia Symptom Checklist (ASKL) forms will be filled.

Patients will be randomly divided into two groups. Patients in the control group will be given beta-blocker therapy, the standard treatment. The local anesthetic agent bupivacaine will be injected into the greater/small occipital nerves and supratrochlear/ supraorbital nerves. Patients in the study group will be asked to keep a diary of pain, dizziness, and painkiller use for one month. At the end of the 1st month, the scoring will be repeated, and the patients who show a decrease in half will be accepted to the next stage, botulinum toxin application. BoNT/A botulinum toxin A (botox; Allergan) will be injected bilaterally into the same regionns. All scoring will be repeated in the 1st, 3rd and 6th months.

ELIGIBILITY:
Inclusion Criteria:

* vestibuler migraine(IHCD3)
* probable vestibular migraine (IHCD3)

Exclusion Criteria:

* Systemic disorders unsuitable for injection administration
* Keloidal scarring
* Neuromuscular disorders
* Botulinum toxin allergies
* Body dysmorphic disorder
* Pregnancy
* Breastfeeding
* Amyotrophic lateralizing sclerosis myopathies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
MIDAS(Migraine Disability Assessment) | 6 months
  The MIDAS (Migraine Disability Assessment) questionnaire is used to measure the impact of headaches. It will be measured at baseline and 6 months after treatment to assess the effects of treatment on vestibular symptoms. Complete recovery will result in significant recovery (>50%), moderate recovery (25-50% reduction), and minimal recovery (<25%).
DHI(Dizziness Handicap Inventory) | 6 months
  The DHI is a 25-item self-report questionnaire that quantifies the impact of dizziness on daily life by measuring self-perceived handicap. It will be measured at baseline and 6 months after treatment to assess the effects of treatment on vestibular symptoms. Complete recovery will result in significant recovery (>50%), moderate recovery (25-50% reduction), and minimal recovery (<25%).
VSS(Vertigo symptom sclae) | 6 months
  The VSS assesses patient-reported symptoms of vestibüler disease. Complete recovery will result in significant recovery (>50%), moderate recovery (25-50% reduction), and minimal recovery (<25%).

SECONDARY OUTCOMES:
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | 6 months
  The relationship between the improvement of vertiginous symptoms and the improvement of psychiatric symptoms will be observed. To evaluate this result, the difference between baseline and post-treatment DASS-21 will be compared
Allodynia Symptom Checklist | 6 months
  The relationship between the improvement of vertiginous symptoms and cutaneous symptoms will be observed. To evaluate this result, the difference between baseline and post-treatment ASCL scores will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Head of Department
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No